CLINICAL TRIAL: NCT07289971
Title: Comparative Evaluation of Clinical and Radiographic Treatment Outcomes of Garlic Gel and Calcium Hydroxide as an Intracanal Medicament in Nonsurgical Root Canal Treatment of Permanent Teeth: A Randomized Controlled Trial.
Brief Title: Comparative Evaluation of Clinical and Radiographic Treatment Outcomes of Garlic Gel and Calcium Hydroxide as an Intracanal Medicament in Nonsurgical Root Canal Treatment of Permanent Teeth.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zara Rizwan, Principal investigator, MDS Resident, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00/220/22
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Apical Periodontitis; Periapical Radiolucency
Keywords: Intracanal Medicament; Allium Sativum; Calcium hydroxide; Root canal treatment; Periapical Index; Resolution of Periapical Radiolucency; Visual Analogue Scale; Palpation; Percussion
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: Double-blinded parallel arm randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group(n=48) (Experimental): Garlic gel will be used as an intracanal medicament
  Interventions: Drug: Allium Sativum as an intracanal medicament
- Control group(n=48) (Active Comparator): Patients will receive informed consent, clinical exam, and preoperative radiographs. After anesthesia and rubber dam isolation, access, cleaning, and shaping of canals will be performed using standard endodontic techniques. Calcium hydroxide (control) will be placed as intracanal medicament, followed by temporary restoration of Cavit and Glass Ionomer cement. After 14 days, if clinical symptoms of pain, tenderness to palpation and percussion resolve, the medicament will be removed, and the canal will be obturated and permanently restored. However, if the patient remains clinically symptomatic, then another dressing of calcium hydroxide will be placed. Finally, clinical outcomes will be recorded after a month and obturation will be delayed until the complete resolution of clinical signs and symptoms. Patients will return after 6 months for clinical and radiographic evaluation, with pre- and postoperative radiographs compared by two endodontists.
  Interventions: Drug: Allium Sativum as an intracanal medicament

INTERVENTIONS:
Drug: Allium Sativum as an intracanal medicament — Patients will receive informed consent, clinical exam, and preoperative radiographs. After anesthesia and rubber dam isolation, access, cleaning, and shaping of canals will be performed using standard endodontic techniques. A sterile paper point will be placed in the canal for pH evaluation, followed by placement of garlic gel with lentulo spiral and temporary restoration of MD Temp and GC Gold Label 2 GIC. Patients will return after 14 days; if symptoms persist, the medicament will be replaced, and the patient will be reviewed again after 14 days and then after one month. Final obturation will only be done once all symptoms have resolved. If the experimental group continues to show symptoms after three dressings, the case will be considered a failure and treated conventionally. When asymptomatic, the medicament will be removed, canals will be irrigated, dried, obturated with gutta-percha and Endoplus sealer. Radiographic outcomes will be evaluated after 6 months by 2 endodontists.

SUMMARY:
Researchers want to check how well garlic works inside permanent teeth as a medicament during root canal treatments. Garlic has shown to possess many helpful properties, like reducing inflammation, helping wounds heal, and antimicrobial characteristics. Because conventional medicaments can be expensive or have potential side effects, researchers are actively exploring natural options like garlic. Some lab studies have already shown that garlic gel can kill the microbes inside the teeth. However, no real-life clinical or X-ray studies have been done on using garlic in permanent teeth. This study may help scientists find a much safer and effective new material for dental treatments in the future.

DETAILED DESCRIPTION:
Clinical trials are needed to evaluate the effectiveness of Allium sativum as an intracanal medicament due to its various useful properties, such as anti-inflammatory, wound healing action, and antimicrobial properties. To overcome the problems with synthetic medicament, researchers are looking for natural alternatives due to their low cost, easy availability, and safety. The objective of the study is to evaluate and compare the clinical and radiographic treatment outcomes of using garlic gel and calcium hydroxide paste as an intracanal medicament in nonsurgical root canal treatment of permanent teeth in terms of:

* Pain.
* Tenderness to palpation.
* Tenderness to percussion.
* Size of Periapical radiolucency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the physical status of ASA I and ASA II according to ASA classification.
* Patients aged from 15-45 years.
* Mature permanent single-rooted teeth with closed apices.
* Patients with clinical signs of symptomatic apical periodontitis (pain, tenderness to palpation, and percussion).
* Patients having radiographic evidence of periapical radiolucency of endodontic origin.
* Patients who have not taken antibiotics for the past 14 days.
* Cooperative patients who show good compliance.

Exclusion Criteria:

* Patients with physical status of ASA III, IV, and V according to ASA classification.
* Teeth with a calcified pulp chamber in periapical radiography.
* Patients who have undergone previous endodontic treatment failure and those with the presence of sinus tract on clinical examination.
* Teeth having advanced periodontal disease, with the basic periodontal examination (BPE) of 3 and 4.
* Presence of internal and external resorption of the root as viewed on the periapical radiograph.
* Presence of vertical root fracture and perforation as viewed on the periapical radiograph

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
CLINICAL AND RADIOGRAPHIC OUTCOMES | Time frame for clinical outcomes: Baseline to 2 weeks Time frame for radiographic outcomes: Baseline to 6 months
  Clinical success will be based on the absence of the following clinical signs and symptoms:
  Pain Tenderness to palpation of adjacent soft tissues Tenderness to percussion of involved tooth Radiographic outcomes will be measured in terms of size of Periapical radiolucency. The Periapical status will be assessed using the periapical index (PAI) scoring system by Orstavik. Each tooth will be assigned one of the Periapical index scores for 5 categories within the scale.
  SCORE POSSIBLE OUTCOME
  1. Normal periapical structure
  2. Small changes in bone structures
  3. Change in bone structure with mineral loss
  4. Periodontitis with well-defined radiolucency
  5. Severe periodontitis with exacerbating features
  Periapical radiolucency will be classified as resolved if the Periapical index score is less than or equal to score of 2.

CONTACTS AND LOCATIONS:
Overall Officials: Zara Rizwan, Bachelors of Dental Surgery, Principal Investigator — University of Health science

IPD SHARING:
Plan to Share IPD: No
Sharing IPD in a way that compromises privacy would violate patient consent agreements and breach significant global privacy laws.

REFERENCES:
- [Result] Faghihi T, Haghgoo R, Taghizade F, Zareiyan M, Mehran M, Ansari G. The clinical and radiographic evaluation of Allium sativum oil (garlic oil) in comparison with mineral trioxide aggregate in primary molar pulpotomy. Dent Res J (Isfahan). 2021 Nov 22;18:100. doi: 10.4103/1735-3327.330881. eCollection 2021. PMID 35003565
- See also: Arruda, M., Neves, M., Diogenes, A., Mdala, I., Guilherme, B., Siqueira, J. and Rôças, I., 2018. Infection control in teeth with apical periodontitis using triple antibiotic solution or calcium hydroxide with chlorhexidine: A Randomized Contro — https://pubmed.ncbi.nlm.nih.gov/30144986/
- Available data/document: Study Protocol: PMID: 35852013 — https://pubmed.ncbi.nlm.nih.gov/35852013/ — https://pubmed.ncbi.nlm.nih.gov/